CLINICAL TRIAL: NCT01012388
Title: Post-Marketing Study of Radiesse® Injectable Dermal Filler for the Treatment of Nasolabial Folds in Persons of Color
Brief Title: Radiesse® Injectable Dermal Filler for the Treatment of Nasolabial Folds in Persons of Color
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1206248
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2009-12-23 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Nasolabial Folds
Keywords: Moderate to severe wrinkles and folds such as nasolabial folds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiesse (Experimental)
  Interventions: Device: Radiesse® Injectable Dermal Filler

INTERVENTIONS:
Device: Radiesse® Injectable Dermal Filler — Calcium hydroxylapatite particles suspected in an aqueous based gel carrier

SUMMARY:
Post marketing study to assess the likelihood of hypertropic scarring, keloid formation and hyper- or hypopigmentation in patients with Fitzpatrick Skin Types IV, V, and VI receiving nasolabial fold treatment with Radiesse® Injectable Dermal Filler

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age.
* Has Fitzpatrick Skin Type IV, V, or VI.
* Understands and accepts the obligation not to receive any other procedures or treatments in the nasolabial fold for 6 months.

Exclusion Criteria:

* Has history of hyper- or hypo-pigmentation in the nasolabial folds, keloid formation, or hypertrophic scarring.
* Has a known bleeding disorder or is receiving drug therapy that could increase the risk of bleeding.
* Has nasolabial folds that are too severe to be corrected in one treatment session.
* Has received any dermal filler or other injections, grafting or surgery in either nasolabial fold.
* Is pregnant, lactating, or not using acceptable contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Los Angeles, California
  - Chevy Chase, Maryland
  - Ypsilanti, Michigan
  - New York, New York
  - Philadelphia, Pennsylvania

REFERENCES:
- [Result] Marmur ES, Taylor SC, Grimes PE, Boyd CM, Porter JP, Yoo JY. Six-month safety results of calcium hydroxylapatite for treatment of nasolabial folds in Fitzpatrick skin types IV to VI. Dermatol Surg. 2009 Oct;35 Suppl 2:1641-5. doi: 10.1111/j.1524-4725.2009.01311.x. Epub 2009 Aug 25. PMID 19708876

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiesse Injectable Dermal Filler: Injectable Dermal Filler - Calcium hydroxylapatite particles suspected in an aqueous based gel carrier for subcutaneous injection for the treatment of nasolabial folds
Period: Overall Study
Arm/Group | Radiesse Injectable Dermal Filler
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 88
  >=65 years | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 52 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Number Participants With Hypertropic Scarring, Keloid Formation, Hyper- or Hypopigmentation in Patients With Fitzpatrick Skin Types IV, V, and VI Receiving Nasolabial Fold Treatment
Description: Skin type IV - Burns minimally, tans moderately and easily, Skin type V - Rarely burns, tans profusely; Skin type VI - Never burns, tans profusely
Time Frame: 3 months
Measure: Number; unit: Participants
Arm/Group | Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 100
Participants | 0

2. Primary Outcome: Number Participants With Hypertropic Scarring, Keloid Formation, Hyper- or Hypopigmentation in Patients With Fitzpatrick Skin Types IV, V, and VI Receiving Nasolabial Fold Treatment
Description: as for outcome 1
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 100
participants | 0

ADVERSE EVENTS:
Arm/Group | Radiesse Injectable Dermal Filler
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 27/100
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiesse Injectable Dermal Filler (N=100)
Redness (Skin and subcutaneous tissue disorders) | 16
Bruising (Skin and subcutaneous tissue disorders) | 7
Swelling (Skin and subcutaneous tissue disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves right to review/comment on manuscript intended for publication/presentation which presents trial data. No manuscripts may be submitted for publication without prior review/comment by Sponsor. Title, right to determine disposition of any copyrights, or copyrightable material, first produced/composed in the performance of this research shall remain with PI, provided that PI grants Sponsor irrevocable right to reproduce/translate/use all such copyrighted material for own purposes.